CLINICAL TRIAL: NCT05409807
Title: Comparison of Classical Ultrasound Guided Method and Combined Wearable Display Technology Method With Ultrasound in Interscalene Nerve Block Applied in Shoulder Surgery
Brief Title: Comparison of Classical Ultrasound Screen and Combined Wearable Display in Interscalene Nerve Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ilker Ital, Assistan Professor Doctor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-TF-AR-II-002
Record Dates: First submitted 2022-05-08; First posted 2022-06-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Nerve Block
Keywords: Interscalene Block; Smart Glasses; Wearable Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic Ultrasound Guided (Experimental): Ultrasound guided interscalene nerve block
  Interventions: Device: Ultrasound guided
- Smart Glasses Assisted (Experimental): Ultrasound guided smart glasses assisted interscalene nerve block
  Interventions: Device: Ultrasound guided smart glasses assisted

INTERVENTIONS:
Device: Ultrasound guided smart glasses assisted — Ultrasound guided smart glasses assisted interscalene nerve block
  Arms: Smart Glasses Assisted
Device: Ultrasound guided — Ultrasound guided interscalene nerve block
  Arms: Classic Ultrasound Guided

SUMMARY:
This study hypothesizes that the use of smart glasses (Head-mounted display Vufine, model VUF-110, Vufine Inc., China)) improves the hand-eye coordination and the first-attempt success rate of ultrasound guided interscalene nerve block. This is a single-center, randomized, controlled study comparing the real-time ultrasound image through smart glasses (intervention group) or the ultrasound machine's monitor (control group) during the interscalene block.

DETAILED DESCRIPTION:
Peripheral nerve blocks, which help patients to recover early after surgery, are performed safely and successfully under ultrasound guidance. Ultrasound-guided peripheral nerve blocks provide sufficient anesthesia for the operation alone or can be applied in combination with general anesthesia and provide postoperative analgesia.

Investigators encounter new developments in health technologies almost every day. With the development of smart technologies and the spread of wearable devices, their use in the field of health is increasing day by day.

Hand-eye coordination is an important skill, especially in the use of ultrasound. The inserted needle should be followed during the procedure in the appropriate area and safely delivered to the desired area.

Patients will be divided into either the study group or the control group. Interscalene nerve block will be performed with preoperative sedation, ultrasound guidance and nerve stimulator.

Interscalene nerve block will be applied to the patients in the study group by using the smart glasses screen, and to the patients in the control group with the conventional ultrasound screen.

In this clinical study, the first trial success rate of the procedures, the time spent during the procedure, the overall success rate, the ergonomics of the practitioner, and the complications related to the block will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to undergo surgery under general anesthesia
* Patients scheduled for postoperative analgesia after shoulder surgery

Exclusion Criteria:

* Local anesthetic allergy
* Skin disease, infection, hematoma
* Chronic obstructive pulmonary disease
* Hepatic, renal, cardiac failures
* Pregnancy
* Uncooperative patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate | During peripheral nerve block procedure. Not to exceed 20 minutes
  Ultrasound visualization and neurostimulator confirmation of the nerve plexus sheath being reached

SECONDARY OUTCOMES:
Overall attempt | During peripheral nerve block procedure. Not to exceed 20 minutes
  Number of attempt of needling
Ultrasound image time | During peripheral nerve block procedure. Not to exceed 20 minutes
  From ultrasound probe application, to get nerves image on the ultrasound screen
Nerve block time | During peripheral nerve block procedure. Not to exceed 20 minutes
  From needle puncture, to local anesthetic spreading
Overall success rate | During peripheral nerve block procedure. Up to 1 day
  The sensory and motor effect of the block
Operator's satisfaction | During peripheral nerve block procedure. Not to exceed 20 minutes
  Operator's satisfaction, 5 scale (Worst, Poor, Acceptable, Good, Best)
Complication rate | Through study completion, an average of 2 week
  Block failure, pneumothorax, hematoma, local anesthetic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Ital, MD, Principal Investigator — Bolu Abant İzzet Baysal Medical School
Locations (1):
- Bolu Abant İzzet Baysal University Faculty of Medicine, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon JW, Richter K, Vivas-Buitrago T, Kim EJ, Chen RE, Quinones-Hinojosa A, Diaz-Gomez JL, Clendenen SR. Technical Feasibility and Safety of Ultrasound-Guided Supraclavicular Nerve Block With Assistance of a Wearable Head-up Display. Reg Anesth Pain Med. 2018 Jul;43(5):559-561. doi: 10.1097/AAP.0000000000000803. No abstract available. PMID 29927851
- [Background] Przkora R, Mora J, Balduyeu P, Meroney M, Vasilopoulos T, Solanki D. Ultrasound-Guided Regional Anesthesia Using a Head-Mounted Video Display: A Randomized Clinical Study. Pain Physician. 2021 Jan;24(1):83-87. PMID 33400431
- [Background] Lim H, Kim MJ, Park JM, Kim KH, Park J, Shin DW, Kim H, Jeon W, Kim H, Kim J. Use of smart glasses for ultrasound-guided peripheral venous access: a randomized controlled pilot study. Clin Exp Emerg Med. 2019 Dec;6(4):356-361. doi: 10.15441/ceem.19.029. Epub 2019 Dec 31. PMID 31910508
- [Background] Jang YE, Cho SA, Ji SH, Kim EH, Lee JH, Kim HS, Kim JT. Smart Glasses for Radial Arterial Catheterization in Pediatric Patients: A Randomized Clinical Trial. Anesthesiology. 2021 Oct 1;135(4):612-620. doi: 10.1097/ALN.0000000000003914. PMID 34352073
- [Background] Kasuya Y, Moriwaki S, Inano C, Fukada T, Komatsu R, Ozaki M. Feasibility of the head-mounted display for ultrasound-guided nerve blocks: a pilot simulator study. J Anesth. 2017 Oct;31(5):782-784. doi: 10.1007/s00540-017-2371-x. Epub 2017 May 5. PMID 28477229